CLINICAL TRIAL: NCT04933799
Title: A Randomized , Double-Blind, Placebo-Controlled, Parallel Group, Phase 2 Trial Assessing the Efficacy and Safety of PF-06650833 in Hospitalized Patients With COVID-19 Pneumonia and Exuberant Inflammation.
Brief Title: IRAK 4 Inhibitor (PF-06650833) in Hospitalized Patients With COVID-19 Pneumonia and Exuberant Inflammation.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Giovanni Franchin, M.D, Ph.D (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Giovanni Franchin, M.D, Ph.D, Study Principal Investigator, Bronx-Lebanon Hospital Center Health Care System
Organization: Bronx-Lebanon Hospital Center Health Care System (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PNA-COV
Record Dates: First submitted 2021-04-23; First posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: COVID-19 Pneumonia
Keywords: COVID-19 Pneumonia; Viral Pneumonia; Pneumonia; COVID-19; COVID; Protein Kinase Inhibitors; Enzyme Inhibitors; Molecular Mechanisms of Pharmacological Action; IRAK 4 Inhibitor; SARS-CoV-2 Pneumonia; IRAK-4 Inhibitor in SARS-CoV-2 Pneumonia
MeSH Terms: conditions — Pneumonia, Viral; Pneumonia; COVID-19 | interventions — 1-(((2S,3S,4S)-3-ethyl-4-fluoro-5-oxopyrrolidin-2-yl)methoxy)-7-methoxyisoquinoline-6-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The research Pharmacists are unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-06650833 + Standard of Care treatment (Active Comparator): Subjects randomized to the PF-06650833 arm of the study will receive 400 mg PF-06650833 (2 x 200 mg tablets) of the MR formulation orally QD under fasted conditions (preferably at least 4 hours after and 1.5 hours before a meal). Subjects who cannot take tablets PO will receive PF-06650833 200 mg IR suspension formulation every 6 hours (NG tube or OG tube, or equivalent). Subjects for whom concomitant administration of a strong inhibitor of CYP3A4 (eg, ritonavir) will have the dose reduced to either 200 mg MR or IR QD. All dosing of study drug will be in addition to current hospital SOC treatment that must include treatment targeting SARS-CoV-2.
  Interventions: Drug: PF-06650833
- Placebo + Standard of Care treatment (Placebo Comparator): Placebo will match the Active comparator in dosage form, dosage, frequency and duration.
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: PF-06650833 — PF-06650833 is an investigational, highly potent and selective, reversible inhibitor of IRAK4. IRAK4 is a serine, threonine kinase that is a key intracellular signaling node downstream of the myddosome-associated Toll-Like Receptors (TLR) 1, 2, 4, 5, 6, 7, 8, 9 and 10, and the interleukin (IL)-1 family receptors (IL-1R, IL-18R and IL-33R) that mediate much of the innate immune signaling.
  As an inhibitor of TLR signaling, PF-06650833 targets a different part of the immune system from the Janus kinase (JAK) inhibitors. Given the partial redundancy of innate immune signaling through IRAK4-independent TLR pathways and the lack of direct suppression of T- and B-cell signaling, PF-06650833 is unlikely to lead to exaggerated immunosuppression.
  Other Names: IRAK 4 inhibitor
  Arms: PF-06650833 + Standard of Care treatment
Drug: Matching Placebo — Placebo will match the study drug in dose, formulation, route and frequency.
  Other Names: Placebo
  Arms: Placebo + Standard of Care treatment

SUMMARY:
The aim of the current clinical study is to evaluate the efficacy and safety of inhibition of Interleukin-1 receptor associated kinase 4 (IRAK4) in ameliorating the proinflammatory state and improving outcomes in severe COVID-19.

DETAILED DESCRIPTION:
Study Design Proposed is a randomized, double-blind, placebo-controlled, parallel group Phase 2 study of the efficacy and safety of PF-06650833, an investigational drug, in hospitalized adult male and female patients with severe COVID-19 and pneumonia, who require supplemental oxygen (O2) support but, who do not need mechanical ventilation or ECMO, to maintain adequate oxygenation.

Patients with confirmed severe acute respiratory syndrome-Coronavirus-2 (SARS-CoV-2) infection, and meeting all other inclusion and exclusion criteria, will be randomized within 3 days of screening to receive PF-06650833 400 mg modified release (MR) tablets (2 x 200 mg tablets) or matching placebo administered orally once daily (QD), under fasted conditions (preferably about 4 hours after and 1.5 before a meal) for up to 28 days (or until discharged from the hospital should this occur earlier). Subjects unable to take tablets by mouth will receive a 200 mg dose of PF-06650833 as an immediate release (IR) suspension or matching placebo administered orally (via nasogastric [NG] or orogastric [OG] tube) every 6 hours, under fasted conditions (as feasible, and preferably about 4 hours after and 1.5 before a meal). Subjects for whom concomitant administration of a strong inhibitor of cytochrome P450 (CYP) 3A4 (eg, ritonavir) will have the dose reduced to either 200 mg MR or IR QD. All dosing of study drug will be in addition to current hospital SOC treatment, that must include some treatment targeting SARS-CoV-2 (eg, remdesivir, if available under emergency use authorization, and/or other targeted anti-viral therapies considered SOC treatment, some of which may also be experimental). Subjects will be assessed daily while hospitalized for a variety of clinical, biomarker, safety, pharmacokinetic (PK), and laboratory parameters.

Number of Study Sites One study site: BronxCare Health System (Bronx Care Hospital; additional site[s] may be added).

Study Population The study population will be derived from patients admitted to the hospital, and will consist of adult male and female patients with severe COVID-19 (pneumonia requiring oxygenation support), aged ≥18, with laboratory-confirmed SARS-CoV-2 infection.

Number of Participants Approximately 68 patients will be recruited to receive PF-06650833 in addition to SOC or placebo plus SOC treatment in a 1:1 ratio. This study utilizes an adaptive design with sample size re-estimation at the interim analysis, with the maximum sample size at 136 subjects.

Outcome Variables

The 8-point National Institute of Allergy and Infectious Diseases (NIAID) ordinal scale of disease severity is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows:

1. Not hospitalized, no limitations on activities.
2. Not hospitalized, limitation on activities and/or requiring home oxygen*.
3. Hospitalized, not requiring supplemental oxygen* - no longer requires ongoing medical care.
4. Hospitalized, not requiring supplemental oxygen* - requiring ongoing medical care (COVID-19 related or otherwise).
5. Hospitalized, requiring supplemental oxygen*.
6. Hospitalized, on non-invasive ventilation or high-flow oxygen devices**.
7. Hospitalized, on invasive mechanical ventilation or ECMO.
8. Death.

   * For subjects on chronic home O2 supplementation (pre-morbid state), supplemental O2 is defined as ≥ home O2 requirement.

     * Use of non-invasive ventilation for chronic conditions (eg, Obstructive sleep apnea [OSA]) is not applicable.

Primary Outcome Variable

• Proportion of subjects worsened at end of treatment (Day 29), as defined by categories 7 and 8 in the 8-point NIAID scale of disease severity.

Secondary Outcome Variables

* Proportion of subjects improved at end of treatment (Day 29), as defined by categories 1, 2, 3, and 4 in the 8-point NIAID ordinal scale of disease severity.
* Proportion of subjects recovered at end of treatment (Day 29), as defined by categories 1, 2, and 3 in the 8-point NIAID ordinal scale of disease severity.
* All-cause mortality at Days 29 and 61, respectively.
* Time to clinical improvement (defined as an at least 1-point decrease on the 8-point NIAID ordinal scale of disease severity).
* Time to worsening (defined as an at least 1-point increase on the 8-point NIAID ordinal scale of disease severity).
* Percentage of subjects in each category of the 8-point NIAID ordinal scale of disease severity at Days 3, 5, 8, 11, 15, 22, and 29.
* Change in the 8-point NIAID ordinal scale of disease severity from Day 1 to Days 3, 5, 8, 11, 15, 22, and 29, as available.
* Proportion of subjects that have required mechanical ventilatory support through Day 29.
* Safety as assessed by reporting of AEs, changes in clinical laboratory parameters (eg, hemoglobin [Hb], white blood cells [WBCs], platelets, hepatic transaminases, serum creatinine [SCr], bilirubin).
* Proportion of subjects alive with resolution of respiratory insufficiency (defined as not requiring supplemental oxygen to maintain oxygen saturation by pulse oximetry [SpO2] >94% while breathing room air) at Days 29 and 61.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized adult male and female patients, including women of childbearing potential, at least 18 years of age, inclusive. Women of childbearing potential must agree to the protocol-specific contraception requirements.
2. Participant (or legally authorized representative) capable of giving signed informed consent.
3. Laboratory-confirmed novel coronavirus (SARS-CoV-2) infection.
4. Evidence of pneumonia assessed by ALL of the following:

   1. Radiographic imaging (eg, chest x-ray, chest computed tomography [CT] scan, etc.); AND
   2. Clinical assessment (evidence of rales/crackles on exam); AND
   3. SpO2 ≤94% on room air.
5. Evidence of increased inflammation as assessed by hsCRP > ULN AND at least ONE of the following being > ULN (as available):

   1. Ferritin;
   2. Procalcitonin;
   3. D-dimer;
   4. Fibrinogen;
   5. LDH;
   6. PT/PTT.

Exclusion Criteria:

1. Other medical condition other than COVID-19 or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study, eg, acute coronary syndrome.
2. Suspected or known active systemic bacterial, viral (except SARS-CoV2 infection) or fungal infections
3. Active herpes zoster infection.
4. Known active or latent tuberculosis (TB) or history of inadequately treated TB.
5. Active hepatitis B or hepatitis C.

   * Patients with positive hepatitis B surface antigen (HBsAg) will be excluded. Patients who are HBsAg negative but hepatitis B core antibody (HBcAb) positive will need a negative hepatitis B virus deoxyribonucleic acid (HBV DNA) to be allowed to enroll in the study; if the HBV DNA is positive, they will be not eligible.
   * Patients with a positive test for hepatitis C virus (hepatitis C virus antibody; HCV Ab) will need a negative hepatitis C virus ribonucleic acid (HCV RNA; or negative HCV Ab test) and normal liver function (as assessed by liver transaminases and bilirubin within protocol-permitted limits, and no other evidence of compromised liver synthetic ability (eg, albumin and coagulation tests within protocol-permitted limits) to be allowed to enroll in the study, provided other eligibility criteria are met.
6. Known history of human immunodeficiency virus (HIV) infection with a detectable viral load or CD4 count <500 cells/mm3 (or patients for whom documentation of viral load or CD4 counts are not available) will be excluded; patients on highly active anti retroviral treatment, undetectable HIV viral load, and CD4 counts ≥500 cells/mm3 would be eligible).
7. Active hematologic cancer.
8. Metastatic or intractable cancer.
9. Pre-existing neurodegenerative disease.
10. Proven bacterial pneumonia, other serious infection, sepsis, and/septic shock.
11. Requirement for mechanical ventilation, or extracorporeal membrane oxygenation.
12. Severe hepatic impairment defined as Child-Pugh Class B or Class C at baseline.
13. Severe renal impairment with an estimated glomerular filtration rate (eGFR) <50 mL/min/1.73 m2.
14. Known history of nephrolithiasis.
15. Severe anemia (Hb <8.0 g/dL).
16. Any of the following abnormal laboratory vales:

    1. Absolute lymphocyte count <500 cells/mm3;
    2. Absolute neutrophil count (ANC) <1500 cells/mm3;
    3. Platelet count <50,000 cells/mm3;
    4. ALT or AST >5X ULN, or total bilirubin >2X ULN, or other evidence of hepatocellular synthetic dysfunction.
17. Any other medical condition or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
18. Prohibited concomitant therapy.
19. Pregnancy (a negative urine or serum pregnancy test is required for inclusion) or breastfeeding.
20. Immunocompromised patients, patients with known immunodeficiencies or taking potent immunosuppressive agents (eg, azathioprine, cyclosporine).
21. Anticipated survival <72 hours as assessed by the Investigator.
22. Participation in other clinical trials of investigational treatments for COVID-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-01-06 (Actual); Primary Completion 2022-03-06 (Estimated); Study Completion 2022-05-06 (Estimated)

PRIMARY OUTCOMES:
Worsening based on the NIAID Ordinal scale | 29 days
  Proportion of subjects worsened at end of treatment (Day 29), as defined by categories 7 and 8 in the 8-point NIAID scale of disease severity.
  1. Not hospitalized, no limitations on activities.
  2. Not hospitalized, limitation on activities and/or requiring home oxygen*.
  3. Hospitalized, not requiring supplemental oxygen* - no longer requires ongoing medical care.
  4. Hospitalized, not requiring supplemental oxygen* - requiring ongoing medical care (COVID-19 related or otherwise).
  5. Hospitalized, requiring supplemental oxygen*.
  6. Hospitalized, on non-invasive ventilation or high-flow oxygen devices**.
  7. Hospitalized, on invasive mechanical ventilation or ECMO.
  8. Death.
     * For subjects on chronic home O2 supplementation (pre-morbid state), supplemental O2 is defined as ≥ home O2 requirement.
       * Use of non-invasive ventilation for chronic conditions (eg, Obstructive sleep apnea [OSA]) is not applicable.

SECONDARY OUTCOMES:
Improvement based on the NIAID Ordinal scale | 29 days
  Proportion of subjects improved at end of treatment (Day 29), as defined by categories 1, 2, 3, and 4 in the 8-point NIAID ordinal scale of disease severity.
Recovered based on the NIAID Ordinal scale | 29 days
  Proportion of subjects recovered at end of treatment (Day 29), as defined by categories 1, 2, and 3 in the 8-point NIAID ordinal scale of disease severity.
mortality | 29 days
  All-cause mortality at Day 29
mortality | 61 days
  All-cause mortality at Days 61
Time to clinical improvement based on the NIAID Ordinal scale | 29 days
  Time to clinical improvement (defined as an at least 1-point decrease on the 8-point NIAID ordinal scale of disease severity).
Time to worsening based on the NIAID Ordinal scale | 29 days
  Time to worsening (defined as an at least 1-point increase on the 8-point NIAID ordinal scale of disease severity)
Percentage of subjects in each category of ordinal scale of disease severity | 29 days
  Percentage of subjects in each category of the 8-point NIAID ordinal scale of disease severity at Days 3, 5, 8, 11, 15, 22, and 29
Change in disease severity based on the NIAID Ordinal scale | 29 days
  Change in the 8-point NIAID ordinal scale of disease severity from Day 1 to Days 3, 5, 8, 11, 15, 22, and 29, as available. Higher score means worsening outcomes.
mechanical ventilatory support | 29 days
  Proportion of subjects that have required mechanical ventilatory support through Day 29.
Safety assessment by reporting of AEs | 29 days
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
subjects alive with resolution of respiratory insufficiency | 29 days
  Proportion of subjects alive with resolution of respiratory insufficiency (defined as not requiring supplemental oxygen to maintain oxygen saturation by pulse oximetry [SpO2] >94% while breathing room air) at Day 29.
subjects alive with resolution of respiratory insufficiency | 61 days
  Proportion of subjects alive with resolution of respiratory insufficiency (defined as not requiring supplemental oxygen to maintain oxygen saturation by pulse oximetry [SpO2] >94% while breathing room air) at Days 61.

OTHER OUTCOMES:
Change from baseline in inflammatory parameters | 29 days
  Change from baseline in inflammatory parameters (eg, high-sensitivity C-reactive protein [hsCRP], procalcitonin, ferritin, D-dimers, lactate dehydrogenase [LDH], fibrinogen, prothrombin time/partial thromboplastin time [PT/PTT], and troponin) in peripheral blood. • Linear mixed effects model that utilizes the longitudinal measurements will be used. The model will include fixed effects for baseline measurements, treatment, visit/time and treatment by visit/time interaction, age group, remdesivir use.
cytokine panel. Units of measurement for all cytokines in the panel is pg/ml | 29 days
  Change from baseline in cytokine panel (interferon[IFN]-gamma, interleukin [IL]-1 Beta , IL 2, IL 4, IL-5, IL-6, IL-8, IL-10, IL-12p70, IL-13, IL-17, tumor necrosis factor alpha [TNF alpha ], IL-2R [sCD25]), as available in peripheral blood.• Linear mixed effects model that utilizes the longitudinal measurements will be used. The model will include fixed effects for baseline measurements, treatment, visit/time and treatment by visit/time interaction, age group, remdesivir use.
SARS-CoV-2 viral load | 29 days
  Change from baseline in SARS-CoV-2 viral load (in nasopharyngeal swabs, blood, and/or saliva), as available
ICU admission | 29 days
  Proportion of subjects that have required ICU admission
mechanical ventilation | 29 days
  Duration (days) of mechanical ventilation.
Ventilator free | 29 days
  Ventilator free days.
Pharmacokinetics of PF-06650833 | 15 days
  Blood samples for analysis of PF-06650833 exposure will be collected at baseline (before the first dose), and at trough before the second dose (if applicable), and at trough on Days 8 and 15, as available.
Pharmacokinetics of PF-06650833 metabolites | 15 days
  Blood samples for analysis of PF-06650833 may be used for determination of metabolites including PF-06787899 and PF 06787900. PF-06650833 may cause the manifestation of atypical, needle-like crystals (that are likely principally precipitates of metabolites of PF-06650833) in urine sediment.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Franchin, M.D, Ph.D, Principal Investigator — Bronx-Lebanon Hospital Center Health Care System
Locations (1):
- Bronx-Lebanon Hospital Center Health Care System, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No